CLINICAL TRIAL: NCT05849324
Title: The Difference of Intravascular Injection Rate During Lumbar Transforaminal Epidural Block Using Bent Needle Compared to Straight Needle: a Prospective Study
Brief Title: Intravascular Injection Rate During Lumbar Transforaminal Epidural Block Using Bent or Straight Needles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Saeyoung Kim, MD, PhD, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2023-03-022-001
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Analgesia, Epidural
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Straight needle (Experimental): 25 gauge straight chiba needle
  Interventions: Device: Straight needle
- Bent needle (Active Comparator): 25 gauge bent chiba needle
  Interventions: Device: Bent needle

INTERVENTIONS:
Device: Straight needle — Lumbar transforaminal epidural steroid injection is a useful option in the diagnosis and treatment of lumbar radicular pain. During lumbar transforaminal epidural steroid injection, straight needle is going to be used.
  Arms: Straight needle
Device: Bent needle — Lumbar transforaminal epidural steroid injection is a useful option in the diagnosis and treatment of lumbar radicular pain. During lumbar transforaminal epidural steroid injection, bent needle is going to be used.
  Arms: Bent needle

SUMMARY:
The primary aim of this study was to compare intravascular injection rates during LTFESI between commonly used straight and bent chiba needles.

DETAILED DESCRIPTION:
Lumbar transforaminal epidural steroid injection (LTFESI) is widely used in clinical practice to effectively deliver injectate into the ventral epidural space. Complications associated with intravascular injection such as spinal cord infarction and paraplegia can occur during LTFESI. The incidence of intravascular injection during LTFESI was known as 9.9% ~ 17.7%. To improve the safety of the procedure, avoidance of intravascular injection is crucial, for which appropriate needle selection is important. Currently, the most commonly used block needles in LTFESI are straight or bent chiba needles.

The primary aim of this study was to compare intravascular injection rates during LTFESI between commonly used straight and bent chiba needles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiating pain from lumbar spinal stenosis and herniated nucleus pulposus.

Exclusion Criteria:

* Pregnancy, allergic to contrast media, patient refusal, and patients with persistent contraindication to nerve block such as coagulopathy and infection of the injection site.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Intravascular injection | During procedure
  Intravascular injection is defined as contrast media spreading out through the vascular channel during injection of contrast media under real time fluoroscopy

SECONDARY OUTCOMES:
Ventral epidural spreading | up to 24 weeks
  Ventral epidural spreading is defined when the contrast reached just behind the vertebral body in fluoroscopic lateral view.
Medial epidural spreading | up to 24 weeks
  Medial epidural spreading is defined as contrast filling the inner side of the pedicle medial margin
Procedure time | During procedure
  Procedure time is defined as the time from the point when the block needle passed through the skin to observation of the complete contrast flow pattern with real time fluoroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Saeyoung Kim, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea